CLINICAL TRIAL: NCT02582047
Title: Immunogenicity and Safety of an Influenza Vaccine Administered Concomitantly With a 13-Valent Pneumococcal Conjugate Vaccine or 23-Valent Polysaccharide Pneumococcal Vaccine in Elderly Patients
Brief Title: Influenza Vaccine and Pneumococcal Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hee Jin Cheong, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INFLUENZAPNEUMO
Record Dates: First submitted 2015-10-05; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Influenza, Human; Pneumococcal Infections
Keywords: influenza vaccine; pneumococcal vaccine; simultaneous vaccination
MeSH Terms: conditions — Influenza, Human; Pneumococcal Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza vaccination with PPV23 (Active Comparator): concomitant vaccination with trivalent inactivated influenza vaccine and 23-valent polysaccharide pneumococcal vaccine
  Interventions: Biological: Influenza vaccination with PPV23
- Influenza vaccination with PCV13 (Active Comparator): concomitant vaccination with trivalent inactivated influenza vaccine and 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: Influenza vaccination with PCV13

INTERVENTIONS:
Biological: Influenza vaccination with PPV23 — GCflu and Pneumovax-23
  Arms: Influenza vaccination with PPV23
Biological: Influenza vaccination with PCV13 — GCflu and Prevenar-13
  Arms: Influenza vaccination with PCV13

SUMMARY:
Previous studies have demonstrated the immunogenicity and safety of the co-administration of the trivalent inactivated influenza vaccine (IIV3) with the polysaccharide pneumococcal vaccine (PPV) or pneumococcal conjugate vaccine (PCV). However, there is no direct comparison study that evaluates the immunogenicity and safety of IIV3 given concomitantly with PCV13 or PPV23 in the elderly. This study is intended to compare the immunogenicity and safety of concomitant administration in the elderly subjects.

DETAILED DESCRIPTION:
During the influenza vaccination period, 224 healthy elderly volunteers randomly received IIV3 given concomitantly with either PCV13 (PCV13+IIV3) or PPV23 (PPV23+IIV3) in a 1:1 ratio. Serum hemagglutination-inhibiting (HI) antibodies for IIV3 were measured at the time of vaccination and 1 month after vaccination. Adverse events were recorded prospectively in a clinical diary during a 7-day period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥65 years who signed the informed consent

Exclusion Criteria:

* Previous pneumococcal vaccine recipients
* Egg allergy
* History of serious adverse event after vaccination
* Any acute disease or infection
* History of neurological symptoms or signs
* Impairment of immune function or immunosuppressant use
* Bleeding diathesis
* Fever (defined as axillary temperature ³38.0°C) within 3 days
* History of Streptococcal pneumoniae infection within the previous 5 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates (A/H1N1, A/H3N2, and B) | Change from baseline titer at 4 weeks
  Seroconversion: a post-vaccination titer ≥1:40 in subjects with a pre-vaccination titer of <1:10 or a ≥4-fold titer increase in subjects with a pre-vaccination titer of ≥1:10

SECONDARY OUTCOMES:
Seroprotection rates (A/H1N1, A/H3N2, and B) | Change from baseline titer at 4 weeks
  Seroprotection rate: percentage of subjects with a post-vaccination titer ≥1:40
GMT folds (A/H1N1, A/H3N2, and B) | Change from baseline titer at 4 weeks
  GMT-fold change: GMT ratio of the post-vaccination titer to pre-vaccination titer

OTHER OUTCOMES:
Frequency and duration of local and systemic adverse events | Monitor using a clinical diary for seven days after vaccination
  the Food and Drug Administration Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jin Cheong, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (2):
- South Korea (2):
  - Korea University Ansan Hospital, Ansan, Kyoungido
  - Hallym University Gangnam Sacred Hospital, Seoul, Seoul